CLINICAL TRIAL: NCT05842759
Title: Avoiding Postinduction Hypotension: the Clinical ZERO-HYPOTENSION Proof-of-concept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-100896-BO-ff
Record Dates: First submitted 2023-03-05; First posted 2023-05-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hypotension; Anesthesia; Hypotension on Induction
Keywords: Hypotension; Low Blood Pressure; Anesthesia Induction; Surgery
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, clinical interventional proof-of-concept study in 120 patients scheduled for elective major non-cardiac surgery at the University Medical Center Hamburg-Eppendorf.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypotension Avoidance Strategy (Other): After the patients' arrival in the induction area, routine anesthetic monitoring (electrocardiography and pulse oximetry) will be established. In all patients, the arterial catheter for continuous intraarterial blood pressure monitoring will be inserted before anesthetic induction (after the insertion site has been infiltrated with a local anesthetic). An uncalibrated pulse wave analysis monitor (MostCareUP, Vygon, Aachen, Germany) will be connected to the patient monitor for advanced hemodynamic monitoring of including cardiac output, systemic vascular resistance, stroke volume variation, and pulse pressure variation.
  Besides continuous intraarterial blood pressure monitoring, the hypotension avoidance strategy will be applied.
  Interventions: Procedure: Monitoring; Procedure: Norepinephrine preparation; Procedure: Propofol administration; Procedure: Alarm adjustment; Procedure: Intervention threshold

INTERVENTIONS:
Procedure: Monitoring — Continuous blood pressure monitoring
Procedure: Norepinephrine preparation — Norepinephrine infusion will be prepared and connected to peripheral or central venous catheter (infusion will not be started)
Procedure: Propofol administration — Propofol infusion will be started only when clinical effects of opioid are noticeable: 1.5 mg/kg propofol in patients less than 55 years old and 1.0 mg/kg propofol in patients 55 years or older over 90 seconds
Procedure: Alarm adjustment — Lower mean arterial pressure alarm threshold will be set to 75 mmHg
Procedure: Intervention threshold — Lower mean arterial pressure intervention threshold will be 75 mmHg: continuous norepinephrine infusion will be started when mean arterial blood decreases below 75 mmHg

SUMMARY:
In this clinical proof-of-concept study, the aim is to investigate the efficacy of a hypotension avoidance strategy to prevent post-induction hypotension. Specifically, it will be investigate how much postinduction hypotension occurs when using a hypotension avoidance strategy - combining continuous intraarterial blood pressure monitoring, careful administration of anesthetic drugs, and continuous administration of norepinephrine to treat hypotension - in high-risk patients having elective non-cardiac surgery.

DETAILED DESCRIPTION:
Hypotension is common in patients having non-cardiac surgery with general anesthesia and is associated with organ injury. About one third of hypotension occurs "postinduction" - i.e., after the induction of general anesthesia but before surgical incision. Unmodifiable risk factors for postinduction hypotension include age, male sex, and a high American Society of Anesthesiologists physical status. However, postinduction hypotension is mainly driven by modifiable factors - specifically, anesthetic drugs that cause vasodilation. Vasodilation can be effectively treated with vasopressors, e.g. norepinephrine.

It is reasonable to assume that postinduction hypotension is largely avoidable by careful anesthetic and hemodynamic monitoring and management during anesthetic induction. A hypotension avoidance strategy could include continuous intraarterial blood pressure monitoring, careful administration of anesthetic drugs, and continuous administration of norepinephrine to treat hypotension. However, it remains unknown to which extent a hypotension avoidance strategy actually can avoid postinduction hypotension. Before testing the effectiveness of hypotension avoidance strategies in large-scale randomized trials it is important to investigate their efficacy.

In this clinical proof-of-concept study, the aim is to investigate the efficacy of a hypotension avoidance strategy to prevent post-induction hypotension. Specifically, it will be investigate how much postinduction hypotension occurs when using a hypotension avoidance strategy - combining continuous intraarterial blood pressure monitoring, careful administration of anesthetic drugs, and continuous administration of norepinephrine to treat hypotension - in high-risk patients having elective non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification III or higher, and in whom intraarterial blood pressure monitoring is planned for clinical indication

Exclusion Criteria:

* Emergency surgery
* Transplant surgery
* History of organ transplant
* Sepsis
* Pregnancy
* Contraindications for the use of propofol
* Rapid sequence induction

Ages: 45 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Area under a MAP of 65 mmHg | First 15 minutes of induction of general anesthesia
  Area under a mean arterial pressure (MAP) of 65 mmHg within the first 15 minutes of anesthetic induction [mmHg x min].

SECONDARY OUTCOMES:
Area under threshold | First 15 minutes of induction of general anesthesia
  Area under a MAP of 60, 50, and 40 mmHg [mmHg x min]
Duration | First 15 minutes of induction of general anesthesia
  Duration of MAP <65, <60, <50, and <40 mmHg [min]
Any Hypotension | First 15 minutes of induction of general anesthesia
  Absolute [n] and relative [%] number of patients with any MAP measurement <65, <60, <50, and <40 mmHg
1-minute Hypotension | First 15 minutes of induction of general anesthesia
  Absolute [n] and relative [%] number of patients with at least one 1-minute episode of a MAP <65, <60, <50, and <40 mmHg
Area above the curve | First 15 minutes of induction of general anesthesia
  Area above a MAP of 100, 110, 120, 140 mmHg [mmHg x min]
Norepinephrine | First 15 minutes of induction of general anesthesia
  Cumulative dose of norepinephrine indexed to body weight [μg kg-1]

OTHER OUTCOMES:
Cardiac Output/Index (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
Stroke Volume/Index (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
dP/dt (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
Eadyn (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
Stroke volume variation (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
Pulse pressure variation (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.
Systemic vascular resistance (Exploratory Endpoint) | First 15 minutes of induction of general anesthesia
  Descriptive analysis including minimum value, duration under threshold, area under threshold, absolute and relative number of patients with at least one episode under threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Flick, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Kristen Thomsen, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No